CLINICAL TRIAL: NCT05887206
Title: Corneal Toxicity in Patients Treated by Belantamab Mafodotin : How to Improve and Facilitate Patients Follow-up Using Refractive Shift ?
Brief Title: Corneal Toxicity in Patients Treated by Belantamab Mafodotin
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN292021/CHUSTE
Record Dates: First submitted 2023-05-17; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Myeloma Multiple
Keywords: Myeloma; relapsed or refractory multiple myeloma (RRMM); Belantamab mafodotin; microcyst-like epithelial changes (MECs); microcyst; corneal toxicity; refractive shift
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated by Belantamab Mafodotin: patients treated by Belantamab Mafodotin with a refractory multiple myeloma and an ophthalmologic follow-up between January 2020 and February 2022 will be included.
  Data will be collected for patients coming from multiple French centers which followed patients treated by Belantamab Mafodotin between January 2020 and February 2022. They will be obtained by contacting centers through an email sent with a secure mail address.
  Interventions: Other: Collection of datas

INTERVENTIONS:
Other: Collection of datas — The collected data are : sex, age, date of first immunotherapy cycle, dose, date of first consultation, objective refraction in spheric equivalent, keratometry, visual acuity, microcyst-like epithelial changes (MECs), location and density, corneal toxicity grade and complementary exams (topography, in vivo confocal microscopy).

SUMMARY:
Belantamab Mafodotin is the first antibody conjugate targeting B-cell maturation antigen (BCMA) in relapsed or refractory multiple myeloma (RRMM). It is used in multiple myeloma refractory to an immunomodulatory drug or proteasome inhibitor and refractory and/or intolerant to an anti-CD38 monoclonal antibody.

It has been found that the immunotherapy causes corneal side effects, Microcyst-like Epithelial Changes (MECs). They are round-shaped corneal inclusions that migrate from the peripheral cornea to the center, causing blurry vision, dryness and refractive shifts depending on their location and density.

DETAILED DESCRIPTION:
This study aims at analysing the refractive shifts caused by Microcyst-like Epithelial Changes (MECs) and whether it can be used to monitor patients and facilitate their follow up.

Constitution of a French multicenter cohort.

ELIGIBILITY:
Inclusion Criteria:

* French patients with a refractory multiple myeloma and an ophthalmologic follow-up between January 2020 and February 2022
* Patients treated by Belantamab Mafodotin

Exclusion Criteria:

* Patients with more than 50% of missing ophthalmologic data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a refractory multiple myeloma, treated by Belantamab Mafodotin, and an ophthalmologic follow-up between January 2020 and February 2022 will be included.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
Keratopathy and Visual Acuity (KVA) scale | Months: 24
  This scale is defined by 4 values : G1, G2, G3 and G4 (the best value is G1)
  The severity grade of microcyst-like epithelial changes (MECs) is rated using the Keratopathy and Visual Acuity (KVA) scale after slit lamp examination.
  The aim is to show a correlation between refractive shift and severity grade of microcyst-like epithelial changes (MECs)
Refraction (no unit) | Months: 24
  The refraction is measured in spheric equivalent (SEQ) with an automated refractometer
  The aim is to show a correlation between refractive shift and severity grade of microcyst-like epithelial changes (MECs)

SECONDARY OUTCOMES:
Monoyer scale | Months: 24
  The score is from 10/10 (best visual acuity) to 1/10 (worth visual acuity) Correlation between visual acuity and severity grade of microcyst-like epithelial changes (MECs)
Parinaud scale | Months: 24
  The score is from 10/10 (best visual acuity) to 1/10 (worth visual acuity) Correlation between visual acuity and severity grade of microcyst-like epithelial changes (MECs)
Keratometry (diopter = 1/m) | Months: 24
  Keratometry is measured in diopter using an autorefractometer or a topograph. This device measures the curvature of the anterior corneal surface based on the power of a reflecting surface. It does this by measuring the size of an image reflected from 2 paracentral points and utilizes doubling prisms to stabilize the image enabling more accurate focusing.
  Correlation between keratometry and severity grade of microcyst-like epithelial changes (MECs)
Epithelial pachymetry (µm) | Months: 24
  Epithelial pachymetry is measured in micrometer (µm) using a topograph
  Correlation between epithelial pachymetry and severity grade of microcyst-like epithelial changes (MECs)

CONTACTS AND LOCATIONS:
Overall Officials: Marie Caroline TRONE, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (10):
- France (10):
  - CHU Dijon, Dijon
  - CHU de Limoges - Hôpital Dupuytren, Limoges
  - HCL- Croix Rousse, Lyon
  - Clinique Monticelli-Vélodrome, Marseille
  - CHRU de Nancy, Nancy
  - CHU Nice, Nice
  - APHP - Kremlin-Bicêtre, Paris
  - CHU Saint-Etienne, Saint-Etienne
  - CHRU Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No